CLINICAL TRIAL: NCT06535074
Title: Differentiating Pathophysiological Mechanisms of Hypoxemia Episodes by Continuous Lung Function Monitoring in Preterm Infants
Brief Title: Lung Function Monitoring During Hypoxemia Episodes
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Deepak Jain. MD, Professor of Pediatrics, Rutgers, The State University of New Jersey
Other Study IDs: Pro2023000655
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Hypoxemia of Newborn
Keywords: electrical impedance tomography; hypoxemia episodes; lung volume

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preterm infants with hypoxemia episodes: Very preterm infants with spontaneous HEs and not receiving invasive mechanical ventilation.
  Interventions: Other: Detecting changes in lung volume with hypoxemia episodes

INTERVENTIONS:
Other: Detecting changes in lung volume with hypoxemia episodes — Electrical impedance tomography (EIT) will be used to assess changes in lung aeration prior and during hypoxemia episodes to classify them into four different subtypes.
  FE subtype: Defined as HEs preceded by reduction in EELI below the baseline.
  Apnea subtype: Defined as HEs not meeting the criteria for FE subtype and preceded by cessation of breathing.
  Mixed subtype: Defined as HEs meeting the criteria for both FE and apnea subtypes.
  Unclassified: Defined as HEs not categorized into any of the above parameters.

SUMMARY:
Premature infants commonly have desaturation episodes due to different reasons such as cessation of breathing or loss of lung volume. The purpose of this study is to differentiate the mechanisms of desaturation episodes with continuous lung volume monitoring. As we better understand the mechanisms underlying the desaturation episodes, newer strategies directed at underlying pathophysiology can potentially by evaluated for mitigation of these episodes.

DETAILED DESCRIPTION:
This is an observational study evaluating changes in lung volume during hypoxemia episodes (HEs or desaturation episodes) in spontaneously breathing very preterm infants. We postulate that HEs can be differentiated into distinct subtypes based on alterations in lung volume. Additionally, the severity and duration of HEs correlates with the degree of changes in lung volumes. Therefore, we are performing an observational study in very preterm infants with spontaneous HEs and classifying these episodes into different subtypes of Apnea, forced exhalation, mixed, and unclassified subtypes according to changes in lung volume. Lung volume will be measured non-invasively using electrical impedance tomography (EIT) device (Sentec Inc, RI, USA). In brief, the device consists of a soft belt with 32 embedded electrodes which is placed around the chest of the infant and applies a weak alternating current and measures returning voltage. The measured returning voltage is dependent on the electrical conductivity of the underlying tissue. The reconstruction algorithm creates an image of regional impedance distribution in real time. These data are then used to compute lung volume parameters at different phases of respiratory cycle providing end expiratory lung impedance reflective of EELV, tidal impedance reflective of tidal volume, and regional distribution of ventilation. The changes in lung volume parameters will be used to differentiate HEs into different subtypes and correlated with degree and severity of HEs. In addition, we will also measure cerebral tissue oxygen saturation (CrSO2) to monitor changes in tissue oxygenation with hypoxemia episodes and changes in lung volume.

ELIGIBILITY:
Inclusion Criteria:

* Born at ≤32w GA
* Post menstrual age between 30w to 36w
* 4 or more episodes of HEs in the previous 24h (Defined as SpO2<90≥5s)

Exclusion Criteria:

* Major congenital malformation
* Receiving invasive mechanical ventilation
* Severe neurological injury
* Hemodynamic instability requiring inotropes in last 72h

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All infants admitted to the neonatal intensive care unit at Bristol Myers Squibb Children's Hospital and meeting eligibility criteria will be considered for enrollment and parents will be approached for informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of hypoxemia episodes of each subtype | 6 hour
  Hypoxemia episodes classified into 4 subtypes of Apnea, forced exhalation, mixed and unclassified according to changes in lung volume parameters.

SECONDARY OUTCOMES:
Frequency of each subtype of episode with severe hypoxemia, prolonged episode, bradycardia | 6hr
  Severe HEs defined as SpO2<80, Prolonged HEs duration>=30s, Bradycardia HR<100 for >=5s
Number of episodes of forced exhalation, apnea not meeting the criteria for hypoxemia episodes | 6hr
  Episodes meeting the EIT criteria for FE and apnea but not associated with HEs
Mean highest change in CrSO2 and cFToE during HEs and each subtype | 6hr
  Change in CrSO2 from baseline and fTOE during HEs

CONTACTS AND LOCATIONS:
Overall Officials: Deepak Jain, MD, Principal Investigator — Rutgers Robert Wood Johnson Medical School Department of Pediatrics
Locations (1):
- Bristol Myers Squibbs Childrens Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and individual patient data meta-analysis.

REFERENCES:
- [Background] Bancalari E, Claure N. Respiratory Instability and Hypoxemia Episodes in Preterm Infants. Am J Perinatol. 2018 May;35(6):534-536. doi: 10.1055/s-0038-1637760. Epub 2018 Apr 25. PMID 29694990
- [Background] Bolivar JM, Gerhardt T, Gonzalez A, Hummler H, Claure N, Everett R, Bancalari E. Mechanisms for episodes of hypoxemia in preterm infants undergoing mechanical ventilation. J Pediatr. 1995 Nov;127(5):767-73. doi: 10.1016/s0022-3476(95)70171-0. PMID 7472834
- [Background] Esquer C, Claure N, D'Ugard C, Wada Y, Bancalari E. Role of abdominal muscles activity on duration and severity of hypoxemia episodes in mechanically ventilated preterm infants. Neonatology. 2007;92(3):182-6. doi: 10.1159/000102056. Epub 2007 Apr 27. PMID 17476118
- [Background] van der Burg PS, Miedema M, de Jongh FH, Frerichs I, van Kaam AH. Cross-sectional changes in lung volume measured by electrical impedance tomography are representative for the whole lung in ventilated preterm infants. Crit Care Med. 2014 Jun;42(6):1524-30. doi: 10.1097/CCM.0000000000000230. PMID 24561568
- [Background] Piraino T. An Introduction to the Clinical Application and Interpretation of Electrical Impedance Tomography. Respir Care. 2022 Jun;67(6):721-729. doi: 10.4187/respcare.09949. PMID 35606004